CLINICAL TRIAL: NCT04943172
Title: The Hancock Jaffe Surgical Antireflux Venous Valve Endoprosthesis (SAVVE) Study
Brief Title: The Hancock Jaffe Surgical Antireflux Venous Valve Endoprosthesis Study
Acronym: SAVVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hancock Jaffe Laboratiores, Inc (Network)
Collaborators: AXIOM Real Time Metrics (Unknown); Syntactx (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P061
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Deep Venous Insufficiency (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- VenoValve (Experimental): Subjects who receive VenoValve implant
  Interventions: Device: Hancock-Jaffe bioprosthetic venous valve (VenoValve®)

INTERVENTIONS:
Device: Hancock-Jaffe bioprosthetic venous valve (VenoValve®) — Surgical implantation of the VenoValve device

SUMMARY:
A prospective, non blinded, single arm, multicenter study designed to assess the safety and effectiveness of the bioprosthetic, VenoValve, which is surgically implanted into the deep venous system for treatment of patients with deep venous valvular insufficiency ( C4b-C6 patients).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the VenoValve System (Hancock Jaffe Laboratories) in human patients. The VenoValve System is designed for treatment of chronic deep venous insufficiency. The VenoValve System enables improvement in chronic lower extremity venous reflux through an open surgical technique. The objective of this study is to assess the safety and effectiveness of the VenoValve System for the treatment of patients with deep venous valvular insufficiency and the associated complications.

ELIGIBILITY:
Inclusion Criteria:

1. Failure of at least 3 months of standard care including compression therapy, and in C6 patients, wound care,
2. Axial deep reflux >1000 msec. at the level of the popliteal vein
3. Venous valvular incompetence from primary or secondary causes, e.g., post-thrombotic syndrome (PTS),
4. CEAP score: C4b, C4c, C5, or C6,
5. Diameter of native target vein ≥8 mm,
6. Age ≥18 years,
7. Ability to tolerate duplex ultrasound,
8. Ability to ambulate without assistance,
9. Able to attend scheduled post-treatment follow-up visits,
10. BMI <40,
11. Willing and able to comply with all compulsory study procedures and provide informed consent prior to any study procedures being performed,
12. Negative COVID-19 test within 6 days of index procedure or record of full vaccination for COVID-19,
13. Female patients of childbearing potential must:

    * have negative pregnancy test at the screening visit or within 7 days of the index procedure, whichever is later,
    * not be breastfeeding or plan to breastfeed through completion of the study,
    * agree to use a medically acceptable method of preventing conception from the screening visit through completion of the study.

Exclusion Criteria:

1. Presence of superficial reflux,
2. Presence of untreated iliac/IVC obstruction greater than 50% in diameter reduction,
3. Previously documented hypercoagulable condition that cannot be adequately treated with anticoagulation,
4. Previous open surgical procedure in the ipsilateral deep venous system,
5. Venous stent in the ipsilateral femoral or popliteal vein,
6. Extensive infrainguinal obstruction of the venous system,
7. DVT or pulmonary embolism within 30 days of the planned procedure,
8. Active malignancy excepting non-melanoma skin cancer,
9. Arterial insufficiency with measured ABI <0.70
10. Lymphedema not due to venous disease,
11. Current or planned participation in another clinical trial within 30 days of treatment,
12. Minor venous procedures (e.g., superficial vein procedures or venous stenting) within 6 weeks of screening,
13. New York Heart Association Class III or greater,
14. Fibromyalgia,
15. Chronic narcotic usage,
16. Positive COVID-19 test within the last 3 months.
17. Other medical conditions or comorbidities which, in the opinion of the investigator, would interfere with study compliance,
18. Contraindication to anticoagulation,
19. Stainless steel sensitivity/ porcine tissue sensitivity,
20. Active superficial thrombophlebitis,
21. Thrombocytosis with platelet count > 1 million/microliter,
22. Unwilling or unable to comply with post-operative anticoagulation regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint is the composite of the following Major Adverse Events: | 30 days
  Death, Major Bleeding, Deep Wound Infection, Ipsilateral deep vein thrombosis, Pulmonary embolism in 75 patients. Rate of >9% is expected

SECONDARY OUTCOMES:
Major Adverse Event rates | 3, 6, 12 months and annually thereafter through 5 years
  Death, Major Bleeding, Deep Wound Infection, Ipsilateral deep vein thrombosis, and Pulmonary Embolism

CONTACTS AND LOCATIONS:
Overall Officials: Marc Glickman, MD, Study Director — Hancock Jaffe Laboratories, Inc
Locations (29):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pima Heart and Vascular, Tucson, Arizona
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - Yale school of Medicine, New Haven, Connecticut
  - Coastal Vascular, Fort Walton Beach, Florida
  - Miami Vascular Specialists, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Saint Louis University, St Louis, Missouri
  - Englewood Health, Englewood, New Jersey
  - Albany Medical Center, Albany, New York
  - Kaleidahealth, Buffalo, New York
  - NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Stony Brook Medicine, New York, New York
  - St. Peter's Vascular Associates, Troy, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - TriHealth, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Jobst Vascular Institute / Promedica Toledo Hospital, Toledo, Ohio
  - UPMC, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Sentara, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ulloa JH, Glickman M. One-Year First-in-Human Success for VenoValve in Treating Patients With Severe Deep Venous Insufficiency. Vasc Endovascular Surg. 2022 Apr;56(3):277-283. doi: 10.1177/15385744211073730. Epub 2022 Feb 7. PMID 35129407